CLINICAL TRIAL: NCT01951456
Title: Resistance Training as an Aid to Smoking Cessation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HL117345-01A1 (NIH)
Record Dates: First submitted 2013-09-10; First posted 2013-09-26 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2018-04

CONDITIONS: Cigarette Smoking
Keywords: Smoking cessation; resistance training
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation | interventions — Resistance Training; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance training (Experimental): Participants will attend two, 45-60-minute progressive, moderate intensity resistance training sessions per week for 12 weeks. The program will maintain a format of a 5-minute warm-up, 35-50 minutes of resistance training and a 5-minute cool-down with flexibility and abdominal exercises.
  Interventions: Behavioral: Resistance training
- Health and Wellness (Active Comparator): Participants in this group will be required to attend the exact same number of sessions as those in the Resistance Training group. Each session will last approximately 45-60 minutes. Sessions will include a practical component/demonstration, an informational video, and a handout on a pertinent healthy lifestyle topic for adults.
  Interventions: Behavioral: Health and Wellness

INTERVENTIONS:
Behavioral: Resistance training
  Arms: Resistance training
Behavioral: Health and Wellness
  Arms: Health and Wellness

SUMMARY:
The purpose of this study is to determine whether resistance training can aid smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

Age 18 or older, smoke five or more cigarettes a day for at least the past 12 months

Exclusion Criteria:

Participating in any type of exercise for >60 minutes/week over the past 3 months, current smokeless tobacco use, participation in an ongoing effort to quit smoking, current or planned pregnancy, any serious medical condition that would make exercise unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-11; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | Change from baseline to 3 months
  Salivary cotinine-verified 7-day Point Prevalence Abstinence (7-day PPA) from nicotine (cigarette smoking).

SECONDARY OUTCOMES:
Cortisol | 3, 6, 12 months
Mood | 3, 6, 12 months
Cigarette cravings | 3, 6, 12 months
Abstinence self-efficacy | 3, 6, 12 months
Sleep | 3, 6, 12 months
Body composition | 3, 6, 12 months
Body weight | 3, 6, 12 months
Lung function | 3, 6, 12 months
Blood pressure | 3, 6, 12 months
Cholesterol profile | 3, 6, 12 months
Glycosylated hemoglobin | 3, 6, 12 months
Muscular strength | 3, 6, 12 months
Aerobic fitness | 3, 6, 12 months
  Six-minute walk test
Smoking cessation | Change from baseline to 6 months
  Salivary cotinine-verified 7-day Point Prevalence Abstinence (7-day PPA) from nicotine (cigarette smoking).
Smoking cessation | Change from baseline to 12 months
  Salivary cotinine-verified 7-day Point Prevalence Abstinence (7-day PPA) from nicotine (cigarette smoking).

CONTACTS AND LOCATIONS:
Locations (1):
- Teachers College, Columbia University, New York, New York, United States